CLINICAL TRIAL: NCT05826171
Title: Priming Motor Learning Through Exercise in People With Spinocerebellar Ataxia: a Randomized Controlled Trial (PRIME-Ataxia RCT)
Brief Title: Priming Motor Learning Through Exercise in People With Spinocerebellar Ataxia
Acronym: PRIME-Ataxia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-088
Record Dates: First submitted 2023-03-22; First posted 2023-04-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6; Spinocerebellar Ataxia Type 7
Keywords: Aerobic Exercise; Balance; Motor Learning; Neurorehabilitation; Telehealth; Spinocerebellar Ataxia; Physical Therapy; Rehabilitation; Cerebellum; High intensity aerobic exercise
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): High-Intensity Aerobic Exercise Prior to Balance Training
  Interventions: Behavioral: High-Intensity Aerobic Exercise Prior to Balance Training
- Group 2 (Active Comparator): Low-Intensity Exercise Prior to Balance Training
  Interventions: Behavioral: Low-Intensity Exercise Prior to Balance Training

INTERVENTIONS:
Behavioral: High-Intensity Aerobic Exercise Prior to Balance Training — 20-30 minutes of high intensity aerobic exercise followed by 20-30 minutes of individualized balance training over telehealth twice weekly, for 8 weeks (16 sessions total). For the aerobic component, participants will be instructed in a 20-30-minute exercise program, using available equipment already located in the participant's home (eg. stationary cycle, elliptical trainer, etc). Exercise intensity is moderate-to-high (between 50-85% Heart Rate Reserve. Participants will be placed on a ramped protocol which increases in intensity slowly over the course of the intervention period. For the balance training component, exercises will consist of steady state, proative, and reactive balance activities that involve sensory integration of vision, proprioception, and vestibular senses. Exercises will be individualized based on baseline assessment outcomes and severity of ataxia as rated by the SARAHome.
  Arms: Group 1
Behavioral: Low-Intensity Exercise Prior to Balance Training — 20-30 minutes of light intensity "warm-up" type exercises, followed by 20-30 minutes of individualized balance training over telehealth twice weekly, for 8 week (16 sessions total). For the "warm-up" exercise component, exercises will consist of stretching and core training. For the balance training component, exercises will consist of steady state, proactive, and reactive balance activities that involve sensory integration of vision, proprioception, and vestibular senses throughout. Exercises will be individualized based on baseline assessment outcomes and severity of ataxia as rated by the SARAHome.
  Both groups are matched for time and frequency of intervention components.
  Arms: Group 2

SUMMARY:
PRIME-Ataxia is a randomized controlled trial that aims to determine the feasibility and efficacy of an 8-week telehealth intervention of high intensity aerobic exercise prior to balance training compared to an 8-week telehealth intervention of low intensity exercise prior to balance training in people with spinocerebellar ataxias (SCAs). The investigators additionally aim to explore changes in motor skill learning on a novel motor skill task in a sub-group of participants pre and post intervention.

DETAILED DESCRIPTION:
The PRIME-Ataxia randomized controlled trial involves 2 groups of participants (n=20). One group (high intensity exercise + balance) will receive high intensity aerobic exercise followed by balance training, and another group (low intensity exercise + balance) will receive low intensity exercise (stretching, warm up exercises) followed by balance training. Both groups will undergo four remote assessments (2 baseline assessments, a mid-intervention assessment, and a post-intervention assessment). A subset of individuals (n=12) from both groups will undergo an in-person assessment on a novel motor task, along with digital posturography assessment of standard functional assessments of mobility and balance at baseline 1 (week 0), and post-intervention (week 16).

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 to 85 years
2. Genetically confirmed diagnosis of SCA1, 2, 3, 6, and 7
3. Scale for Ataxia Rating and Assessment (SARA) score between 8-25/40, capturing mild-moderate disease
4. Able to walk with/without assistive device
5. Successful completion of Physical Activity Readiness Questionnaire (PAR-Q) to confirm no medical contraindications to exercise
6. Care partner availability during assessments and/or intervention pending balance scores

Exclusion Criteria:

1. Severe non-ataxic motor symptoms such as dystonia, tremor, or Parkinsonism, measured by Inventory of Non-Ataxia Signs (INAS)
2. Peripheral sensory loss (as confirmed with monofilament or clinical proprioceptive testing)
3. Severe visual complications associated with ataxia (i.e., Spontaneous nystagmus, retinal or optic nerve involvement, especially in SCA7) defined as as have a score on the Snellen Visual Acuity test = 20/200 - 20/400, OR a visual field of 20 degrees of less.
4. Musculoskeletal injury that would prevent participation in an exercise program
5. Other concurrent disease of the cerebellum (e.g. stroke, multiple sclerosis)
6. Cardiac/pulmonary conditions that would affect participants ability to participate exercise program
7. Currently engaged in >3 week moderate-high intensity aerobic exercise and/or balance training

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Scale for Assessment and Rating for Ataxia | Baseline, Post-Intervention (4 months)
  Clinical rating scale for severity of ataxia symptoms. This is an 8-item clinical performance based scale, which individuals are graded according to total ataxia severity. Total scores can range from 0 (no ataxia) to 40 (most severe ataxia). Scores are based on performance of the following tasks: 1) Gait, 2) Stance, 3), Sitting, 4) Speech Disturbance, 5) Finger Chase, 6) Nose-Finger Test, 7) Fast alternating hand movements, 8) Heel-shin slide. For the purpose of this study, we will be performing a validated modified version of the SARA, referred to as the SARAHome. The SARAHome is comprised of the first four items and item 6 from the original SARA Scale (Gait, Stance, Walking, Speech, and Nose-Finger Test) and it will be administered via telehealth.
Change in Cerebellar Cognitive Affective Syndrome Scale | Baseline, Post-Intervention (4 months)
  The Cerebellar Cognitive Affective Syndrome Scale (CCAS) was developed as a bedside quick screen for Cerebellar Cognitive Affective Symptom (also referred to as Schmalmann's Syndrome). The CCAS is a 10-item scale of cognitive and neuropsychiatric tests detailing executive function, working and verbal memory, language, visuospatial function, abstract reasoning, behavior and affect. Two scores are reported; a raw score ranging from 0 (severe cognitive impairment) to 120 points (no cognitive impairment), as well as a Pass/Fail marker for each of the 10 items on the scale. 1 fail is considered as possible cerebellar cognitive affective symptom, 2 fails are considered probable, and 3 fails are considered clinically definite.
Change in Patient Reported Outcome Measure for Ataxia | Baseline, Post-Intervention (4 months)
  Patient reported outcome measure for people with ataxia. The test was developed to assess 3 domains (physical, activities of daily living, mental health) and 14 subdomains. It has been proven to be valid and reliable against measures of motor ataxia, mental health, and quality of life. The original Patient Reported Outcome Measure for Ataxia has 70 questions, and records a total score out of 280 possible points. For the purpose of this trial, we will use the Short-Form version of this assessment which asks 10 questions, and it scored out of a total of 40 possible points.

SECONDARY OUTCOMES:
Activities Specific Balance Scale (ABC) | Baseline, Post-Intervention (4 months)
  Patient reported outcome evaluating the balance confidence of a participant in performing a variety of activities without losing balance or experiencing a state of unsteadiness. Participants are asked to rank their perceived balance confidence on a scale of 0% (no balance confidence) to 100% (high balance confidence). All scores are summed, and averaged for a total overall estimate of balance confidence.
Digital Biomarker of Static Posturography | Baseline, Post-Intervention (4 months)
  Participant will perform a series of static standing postures and postural sway will be recorded with a smart phone app, and/or inertial measurement units. Measure of postural sway will be recorded (higher values are worse outcomes).
Digital Biomarker of Dynamic Posturography | Baseline, Post-Intervention (4 months)
  Participant will perform a walking test which will be recorded with a smart phone app, and/or inertial measurement units. Measure of postural sway will be recorded (higher values are worse outcomes).
Motor Adaptation | Baseline, Post-Intervention (4 months)
  Prism Adaptation with finger targeting to touchscreen. Performed in a sub-set of participants for this trial.
Neurological Quality of Life | Baseline, Post-Intervention (4 months)
  Self report of health related quality of life for people with neurological conditions. The measure that will be used in this trial is a short-form assessing social or functional roles and abilities. 8 questions with 5-item Likert response, higher score is better outcome.
Patient Global Impression of Change | Baseline, Post-Intervention (4 months)
  Self-report measure that assesses a participants thoughts or beliefs about the efficacy of treatment. The Patient Global Impression of Change scale is a 7 point scale depicting a patient's rating of overall improvement, score 1-7, higher score is better.
Acceptability Questionnaire | Baseline, Post-Intervention (4 months)
  Short open-ended questionnaire to assess the acceptability of the intervention. These open-ended questions will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Quinn, PT, EdD, Principal Investigator — Teachers College, Columbia University; Chelsea E Macpherson, DPT, Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macpherson CE, Awad F, Rana V, Kuo SH, Quinn L. Fatigue Limits Motor and Cognitive Improvements after High-intensity Exercise Prior to Balance Training over Telehealth in People with Spinocerebellar Ataxia. Int J Telerehabil. 2025 Dec 12;17(2):6713. doi: 10.63144/ijt.2025.6713. eCollection 2025. PMID 41445681